CLINICAL TRIAL: NCT05947630
Title: IMPression 3D & ACcès à la Teléréadaptation / 3D-printen en Toegang Tot Telerevalidatie
Brief Title: 3D-printing and Acces to Tele Rehabilitation
Acronym: Imp&acte3D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lieven De Maesschalck (Other)
Collaborators: Handicap International (Other)
Responsible Party: Sponsor-Investigator, Lieven De Maesschalck, Innovation Manager, Thomas More Kempen
Organization: Thomas More Kempen (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: S65004
Record Dates: First submitted 2021-10-07; First posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Orthopedic Disorder
Keywords: lower limb
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- AFO (ankle foot orthosis) dynamic and correctional (Experimental): Groep A with AFO (ankle foot orthosis) dynamic and correctional
  Interventions: Device: Ankle Foot Orthosis (AFO)
- AFO or KAFO (knee ankle foot orthosis) correctional (No Intervention): Groep B with AFO or KAFO (knee ankle foot orthosis) and only correctional
- KAFO dynamic and correctional (Experimental): Groep C with KAFO dynamic and correctional
  Interventions: Device: Knee Ankle Foot Orthosis (KAFO)
- KAFO correctional (No Intervention): Groep D with KAFO only correctional

INTERVENTIONS:
Device: Ankle Foot Orthosis (AFO) — 3D treatment (AFO will be printed) versus traditional made AFO
  Arms: AFO (ankle foot orthosis) dynamic and correctional
Device: Knee Ankle Foot Orthosis (KAFO) — 3D treatment (KAFO will be printed) versus traditional made KAFO
  Arms: KAFO dynamic and correctional

SUMMARY:
This study will investigate whether 3D printing of orthoses (night splints and AFO/KAFO for walking, further named as dynamic AFO/KAFO) for the lower limbs can help to improve the limited accessibility to orthopaedic devices in developing countries. The 3D printed orthoses will be assessed for effectiveness, cost and feasibility. Measurement and manufacture of the orthoses is also supported remotely via video conferencing.

DETAILED DESCRIPTION:
Specifically, the study is being conducted in 3 West African countries: Togo, Niger and Mali. A total of 4 orthopaedic centres are involved, whereby an equal number of patients are recruited everywhere.

There are 2 groups of patients, those who need a (knee) ankle-foot orthosis to move around (dynamic AFO/KAFO) and those who need a night splint to correct the ankle or knee position. All patients in the study will have a treatment route involving fitting a new traditional orthosis and a new 3D printed orthosis. The order of application of both treatments will be randomised in a crossover design. Patients will be measured at baseline after the first treatment period (3 weeks) and after the second treatment period (6 weeks). The primary outcome measures are different for both groups of patients: the walking speed when performing the 10-metre walk test in the patients wearing the dynamic AFO/KAFO, and the measured angle (of knee or ankle) in the patients wearing a night splint.

ELIGIBILITY:
Inclusion Criteria:

* Pathology: foot stance abnormality
* Both unilateral and bilateral orthoses are included
* Pathology: genu varum

Exclusion Criteria:

* Patient is already wearing a night splint
* The patient cannot stand upright
* The patient is pregnant

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2019-04-15 (Actual)

PRIMARY OUTCOMES:
10 meter walk test | 5 weeks
  10 meter walk test
knee angle test | 5 weeks
  Knee angle test
Ankle angle test | 5 weeks
  Ankle angle test

SECONDARY OUTCOMES:
OPUS questionnnaire | 5 weeks
  OPUS questionnnaire (measure on 5 point Likertscale: Very easy, Easy, Slightly difficult, Very difficult and Cannot do this activity and this for 21 items.
Range of motion | 5 weeks
  Range of motion

CONTACTS AND LOCATIONS:
Locations (4):
- CNAOM, Bamako, Mali
- Centre Hospitalier Universitaire de Niamey, Niamey, Niger
- Togo (2):
  - CRAO, Dapaong
  - CNAO, Lomé

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Creylman V, Knippels I, Janssen P, Biesbrouck E, Lechler K, Peeraer L. Assessment of transfemoral amputees using a passive microprocessor-controlled knee versus an active powered microprocessor-controlled knee for level walking. Biomed Eng Online. 2016 Dec 19;15(Suppl 3):142. doi: 10.1186/s12938-016-0287-6. PMID 28105945

DOCUMENTS (2):
  • Study Protocol (2018-05-03): https://cdn.clinicaltrials.gov/large-docs/30/NCT05947630/Prot_000.pdf
  • Informed Consent Form (2018-05-03): https://cdn.clinicaltrials.gov/large-docs/30/NCT05947630/ICF_001.pdf